CLINICAL TRIAL: NCT01247168
Title: An Open-Label, Dose-Escalation Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics fo the PARP Inhibitor AZD2461 in Patients With Refractory Solid Tumors
Brief Title: An Open-Label, Dose-Escalation Study of AZD2461
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3660C00001
Record Dates: First submitted 2010-11-08; First posted 2010-11-24 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Refractory Solid Tumors; Cancer Tumor
Keywords: Refractory; Solid tumors; Cancer
MeSH Terms: conditions — Neoplasms | interventions — AZD2461

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD2461

INTERVENTIONS:
Drug: AZD2461 — oral capsules, continuous dosing and intermittent dosing

SUMMARY:
This study is being conducted to test study drug AZD2461 to see how it may work to treat solid tumors. The main purpose of this study is to determine the safety and tolerability of AZD2461. This is the first time the drug has been given to humans and is classed as a first time in man study. Its main purpose is to establish a safe dosage of the drug and provide additional information on any potential side effects this drug may cause. The study will also assess the blood levels and action of AZD2461 in the body over a period of time and will indicate whether the drug has a therapeutic effect on solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of solid tumor malignancy that is not responsive to standard therapies or for which there is no effective therapy.
* Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1
* Patients must be 18 years of age
* Using adequate contraceptive measures, be surgically sterile or post-menopausal
* Patients entering this study must be willing to provide tissue from a previous tumor biopsy (if available) for correlative testing. If tissue is not available, a patient will still be eligible for enrollment into the study..

Exclusion Criteria:

* Patients currently receiving cancer therapy
* Use of investigation anti-cancer drug or major surgery, radiotherapy or immunotherapy with the last 21 days
* cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of AZD 2461 by collection of adverse events, hematology, clinical chemistry data and vital signs. | Day 1
To determine the maximum tolerated dose of AZD 2461 by collection of adverse events, hematology, clinical chemistry data and vital signs. | Day 8
To determine the maximum tolerated dose of AZD 2461 by collection of adverse events, hematology, clinical chemistry data and vital signs. | every 3 weeks after day 8

SECONDARY OUTCOMES:
To characterize the pharmacokinetic profile of AZD2461 by collection of blood samples for the measurement of AZD2461 in plasma concentration | Continuous dosing Cycle 1 and 2, Day 1 (pre-dose, 1-hr, 6-hr and 24-hr)
To characterize the pharmacokinetic profile of AZD2461 by collection of blood samples for the measurement of AZD2461 in plasma concentration | Intermittent dosing Cycle 1, Day 1 and Day 14 (pre-dose, 1-hr, 6 hr and 24-hr) Day 18 (+/- 2 days) Cycle 2, Day 1 (pre-dose)
evaluate the pharmacodynamic response after treatment with AZD2461 as the change in PARP (Poly (ADP-ribose) polymerase) inhibition in PBMCs (peripheral blood mononuclear cell) | weekly
To explore the clinical tumor response after treatment with AZD2461 as the assessment of patients with overall tumor response Complete Response (CR), Partial Response (PR), duration of response, stable disease (SD) and time to disease progression | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hughes, MA, MB, ChB, PhD, P, Study Director — AstraZeneca; Dr. Jeffrey Infante, MD, Principal Investigator — Sarah Cannon Research Institute (SCRI)
Locations (1):
- Research Site, Nashville, Tennessee, United States